CLINICAL TRIAL: NCT07212543
Title: The Effects of Different Low-Flow Desflurane Anesthesia Strategies on Bispectral Index and Postoperative Cognitive Functions in Patients Undergoing Major Abdominal Surgery
Brief Title: Low-Flow Desflurane Anesthesia and Its Effects on BIS and Postoperative Cognitive Functions
Status: Active, not recruiting | Type: Observational
Sponsor: Dolunay ARIK (Other)
Responsible Party: Sponsor-Investigator, Dolunay ARIK, Resident Doctor (Anesthesiology), Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Organization: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Other Study IDs: 2025-05/73
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Major Abdominal Surgeries
Keywords: Low-flow anesthesia.; Desflurane; Major abdominal surgery; Bispectral Index (BIS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1 :desflurane 0.5 L/min Group 2 :desflurane 1 L/min Group 3 : desflurane 1.5 L/min: This cohort includes adult patients undergoing major abdominal surgery whose general anesthesia is maintained with desflurane using different low-flow strategies. The main intervention of interest is the variation in fresh gas flow rates. Participants will be divided into three subgroups according to the applied flow rate:
  0.5 L/min desflurane anesthesia 1.0 L/min desflurane anesthesia 1.5 L/min desflurane anesthesia During surgery, the depth of anesthesia will be continuously monitored using the Bispectral Index (BIS). Cognitive function will be assessed both preoperatively and postoperatively with the Mini-Mental State Examination (MMSE). This design will allow comparison of the effects of different low-flow strategies on intraoperative BIS values as well as on cognitive function changes before and after surgery.
  Interventions: Other: Routine anesthesia care (desflurane at different low-flow rates: 0.5, 1.0, 1.5 L/min); no intervention assigned as part of the study.

INTERVENTIONS:
Other: Routine anesthesia care (desflurane at different low-flow rates: 0.5, 1.0, 1.5 L/min); no intervention assigned as part of the study. — Routine anesthesia care (desflurane at different low-flow rates: 0.5, 1.0, 1.5 L/min); no intervention assigned as part of the study.

SUMMARY:
This study investigates the effects of low-flow desflurane anesthesia in adult patients undergoing major abdominal surgery. The researchers will examine whether different low-flow strategies:

Cause differences in the Bispectral Index (BIS), which measures brain activity during anesthesia, Affect postoperative cognitive functions such as memory and attention.

Participants will:

Receive desflurane anesthesia during surgery, Have anesthesia delivered at different low-flow rates, Have their BIS values monitored throughout the operation, Complete tests after surgery to evaluate their cognitive functions.

This research will help determine the safety of different low-flow strategies and their impact on patients' cognitive recovery after surgery.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate the effects of different low-flow desflurane anesthesia strategies on intraoperative anesthetic depth, measured by the Bispectral Index (BIS), and on postoperative cognitive functions in patients undergoing major abdominal surgery.

Patients will receive desflurane anesthesia delivered at different low-flow rates. Throughout surgery, BIS values will be continuously monitored to assess the depth of anesthesia. Postoperatively, standardized cognitive function tests will be performed at predetermined time points to evaluate potential cognitive impairment or recovery. The study aims to clarify whether the choice of low-flow strategy influences short-term postoperative neurocognitive outcomes.

Quality assurance and data management procedures:

Data collection will be conducted using standardized electronic case report forms (eCRFs).

All collected data will undergo range and consistency checks against predefined rules.

Source data verification will be performed through comparison with medical records and anesthetic monitoring logs.

A data dictionary will be maintained, documenting each variable, coding standards (e.g., MedDRA where applicable), and reference ranges.

Missing data will be handled according to a predefined plan, with cases flagged as missing, unusable, or inconsistent.

Sample size and statistical plan:

The sample size has been estimated to ensure sufficient statistical power to detect clinically meaningful differences in BIS and postoperative cognitive function scores between different low-flow strategies. Statistical analyses will include descriptive statistics, group comparisons using parametric or non-parametric tests, and regression models where appropriate. A detailed statistical analysis plan has been developed to address both primary and secondary endpoints.

This study will provide evidence regarding the safety and neurocognitive impact of different low-flow desflurane strategies. Findings are expected to support clinical decision-making in optimizing anesthetic management for patients undergoing major abdominal procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-75 years

ASA physical status I-III

Scheduled for elective major abdominal surgery

Provided written informed consent

Normal preoperative neurocognitive function

Exclusion Criteria:

History of neurological or psychiatric disorders

History of cognitive impairment

Diagnosed hepatic or renal insufficiency

Presence of other systemic diseases contraindicating anesthesia

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from patients undergoing elective major abdominal surgery at the Department of Anesthesiology and Reanimation, Ankara Dr Abdurrahman Yurtaslan Onkology Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Mini-Mental State Examination (MMSE) Score Postoperatively | From baseline (preoperative assessment, within 24 hours before surgery) to postoperative assessments at 24 hours and 7 days after surgery
  Measure: Change in cognitive function assessed by the Mini-Mental State Examination (MMSE)
  Time Frame: From baseline (preoperative assessment) to postoperative assessment (within 24 hours after surgery)
  Description: The MMSE will be used to evaluate changes in cognitive function in patients receiving desflurane anesthesia at different low-flow rates. The primary endpoint is the difference between preoperative and postoperative MMSE scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, YENİMAHALLE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bingol Tanriverdi T, Tercan M, Gusun Halitoglu A, Kaya A, Patmano G. Comparison of the Effects of Low-flow and Normal-flow Desflurane Anaesthesia on Inflammatory Parameters in Patients Undergoing Laparoscopic Cholecystectomy. Turk J Anaesthesiol Reanim. 2021 Feb;49(1):18-24. doi: 10.5152/TJAR.2020.30. Epub 2020 Nov 30. PMID 33718901
- [Background] https://www.researchgate.net/publication/319617159_Low_flow_anesthesia_will_gain_eras_enhanced_recovery_after_surgery
- [Background] Baum JA. Low-flow anesthesia: theory, practice, technical preconditions, advantages, and foreign gas accumulation. J Anesth. 1999;13(3):166-74. doi: 10.1007/s005400050050. No abstract available. PMID 14530937